CLINICAL TRIAL: NCT03061396
Title: The Different Effectiveness of Single Acupoint vs Matching Acupoints in Chemotherapy-induced Nausea and Vomiting：A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: The Comparative Study on the Efficacy and Safety of Single Acupoint and Matching Acupoints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: National Basic Research Program, China (Other); West China Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Gansu Provincial Cancer Hospital (Unknown); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Guo, Professor, Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014CB543201-03
Record Dates: First submitted 2017-02-05; First posted 2017-02-23 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Electro-acupuncture; Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture Single point (Experimental): Single point PC6 means there is only one acupoint to be chosen: Neiguan(PC6)
  Interventions: Other: Single points PC6
- Electroacupuncture Matching points (Experimental): There are three acupoints to be chosen:Bilateral Neiguan(PC6)and Zhongwan(CV12)
  Interventions: Other: Matching points PC6+CV12

INTERVENTIONS:
Other: Matching points PC6+CV12 — Choose both Neiguan(PC6) and Zhongwan point(CV12).The needles are connected through a electro-acupuncture apparatus, the positive poles are linked to the needle, and the reference poles are located near the acupoint about 1cm with a electrode.Frequency is 2/10 hertz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10 milliampere. And plus 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron, Tropisetron，Granisetron or Ondansetron) and dexamethasone.
  Arms: Electroacupuncture Matching points
Other: Single points PC6 — Choose Neiguan(PC6)of double upper limb.The needles are connected through a electro-acupuncture apparatus, the positive poles are linked to the needle, and the reference poles are located near the acupoint about 1cm with a electrode.Frequency is 2/10 hertz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10 milliampere. And plus 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron, Tropisetron，Granisetron or Ondansetron) and dexamethasone.
  Arms: Electroacupuncture Single point

SUMMARY:
The purpose of this study is to clarify whether the matching acupoints are more effective than a single point by electro-acupuncture in the management of chemotherapy-induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed as cancer and need to accept chemotherapy
2. The score of Karnofsky ≥70
3. Patients of either gender and age 18 years to 80 years
4. Patients receiving chemotherapy both outpatients and inpatients
5. Patients receiving chemotherapy regime with high risk of causing vomiting: cisplatin ≥60 mg/m2, or joint chemotherapy regime of Anthracyclines (Adriamycin≥ 40 mg/ m2 or epirubicin≥60 mg/m2), Dacarbazine or Carboplatin（area under the curve greater than 5mg/ml/min）
6. Life expectancy > 6 months

Exclusion Criteria:

1. To receive radiotherapy and chemotherapy
2. Gastrointestinal tumors
3. Patients with serious liver disease or abnormal hepatorenal function (Aspartate Aminotransferase, Alanine Aminotransferase , and Total Bilirubin are 3 times more than normal, blood urea nitrogen and Cr are 2 times more than normal)
4. Presence of cardiac pacemaker
5. Inflammatory skin reaction
6. Nausea and/or vomiting resulting from opioids or metabolic imbalance (electrolytic disturbances)
7. Patients unable to provide self-care or communication
8. Nausea and/or vomiting resulting from mechanical risk factors (i.e.,intestinal obstruction)
9. Patients with brain metastases or symptoms of intracranial hypertension
10. Nausea and/or vomiting resulting from other diseases(i.e.,sympathetic cervical dispositions, Meniere's syndrome)
11. Women in pregnant and lactating period
12. Refusal to sign informed consent, rejection of randomization into intervention groups.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-04-28 (Estimated); Study Completion 2018-05-28 (Estimated)

PRIMARY OUTCOMES:
Complete Control rates of Nausea and Vomiting | 6weeks
  There is no emetic episodes, no rescue therapy, and no significant nausea from first day of antiemetic therapy to 5th day.
Complete Response rates of Vomiting | 6weeks
  There is no emetic episodes and no rescue therapy on first day of antiemetic therapy and second day to 5th day.
Nausea and Vomiting visual analogic scale (VAS) | 6weeks

SECONDARY OUTCOMES:
Tcm Gastro-intestinal evaluation | 3weeks
the grading of constipation ,diarrhea and decrease in appetite | 3weeks
  Number of participants with constipation ,diarrhea and decrease events as assessed by CTCAE v4.0
Electrogastrogram | 3weeks
Hospital Anxiety and Depression Scale | 3weeks
Functional Assessment of Cancer Treatment - General scale4.0 | 3weeks

OTHER OUTCOMES:
Number of Participants With Abnormal Laboratory Values | 6weeks
  the number of blood cells,serumAlanine aminotransferase,Aspertate，Aminotransferase,total bilirubin,Creatinine，blood sodium，blood potassium
cardial electrical activity | 6weeks
other adverse effect during the chemotherapy | 6weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of TCM, Tianjin, Tianjin Municipality, China